CLINICAL TRIAL: NCT05182398
Title: Investigation of Validity and Reliability of the Modified Four Square Step Test in Multiple Sclerosis Patients
Brief Title: Validity and Reliability of the Modified Four Square Step Test in Multiple Sclerosis Patients
Status: Withdrawn | Type: Observational
Why Stopped: The study was stopped because the validity and reliability study of the test method was published in the same patient group.
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof., Kahramanmaras Sutcu Imam University
Other Study IDs: ipekkatircikirmaci
Record Dates: First submitted 2021-12-15; First posted 2022-01-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Fall; Modified Four Square Step Test; Multiple sclerosis; Balance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis patient: First day, first evaluator will perform all tests, and second day, second evaluator will perform Modified Four Square Step Test.
  Interventions: Other: Assesment

INTERVENTIONS:
Other: Assesment — Modified Four Square Step Test, Berg Balance Scale, Dynamic Gait Index ,Activity-Specific Balance Confidence Scale

SUMMARY:
Balance disorder is common in people with MS. As the disease worsens, it is associated with impaired balance, difficulty walking, decreased mobility, and an increased risk of falling. Given the prevalence and clinical significance of balance dysfunction in individuals with MS, the assessment of balance has become an important focus in MS clinical practice and research. The Four Square Step Test is a standard clinical measure used to assess dynamic standing balance. It is a timed test in which the individual is instructed to step rapidly forward, backward, and to the right and left over a low obstacle (a cane). The test assesses the ability to quickly change direction of movement and is a timed test involving the use of assistive devices.

In the modified four-square stepping test, the floor is divided into four equal squares with tape instead of a cane. Performing the test with tape, instead of patients at risk of being stuck with a cane, will ensure its applicability to a wider patient population.

The aim of the study is to examine the validity and reliability of the modified four-frame stepping test in MS patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a progressive disease of the central nervous system characterized by demyelination and destruction of motor and sensory axons. As the disease worsens, it is associated with impaired balance, difficulty walking, decreased mobility, and an increased risk of falling. The prevalence of balance dysfunction in individuals with MS and Given its clinical relevance, the assessment of balance has become an important focus in MS clinical practice and research.The Four Square Step Test is a standard clinical measure used to assess dynamic standing balance.The individual rapidly forwards over a low obstacle (a cane), is a timed test in which instructed to step backward and to the right and left.The four-frame stepping test was developed to document deficiencies in stance balance, predict falls, assess self-perceived limitations in walking, and compare changes in standing balance following exercise training. Compared to other standardized tests, scoring is not dependent on the subjectivity of the examiner, can be administered by a person with minimal training, and requires minimal time, space, and equipment. In the modified four-square stepping test, the floor is divided into four equal squares with tape instead of a cane. Performing the test with tape, instead of patients at risk of being stuck with a cane, will ensure its applicability to a wider patient population.

ELIGIBILITY:
Inclusion Criteria:

* Having an EDSS score of 4 and below,
* Being between the ages of 18-65
* Willingness to participate in the study

Exclusion Criteria:

* Being pregnant or within the first 3 months after giving birth,
* Receiving corticosteroid therapy in the last 1 month,
* Using drugs that will affect walking in the last 1 month

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Modified Four Square Step Test | First day
  The square drawn on the floor is divided by tape into 4 equal parts. The number 1 is written in the lower right corner, and the number 4 is written clockwise. With the start command, individuals are asked to step on the numbers in order. First of all, he is asked to take a step forward (to the number 1 and 2), then to the left (to the number 3), then to the back (to the number 4). Then he is asked to take steps from 4 to 1 again. Time is saved
Modified Four Square Step Test | second day
  The square drawn on the floor is divided by tape into 4 equal parts. The number 1 is written in the lower right corner, and the number 4 is written clockwise. With the start command, individuals are asked to step on the numbers in order. First of all, he is asked to take a step forward (to the number 1 and 2), then to the left (to the number 3), then to the back (to the number 4). Then he is asked to take steps from 4 to 1 again. Time is saved

SECONDARY OUTCOMES:
Berg Balance scale | First day
  It is a 14-item scale that measures the ability to maintain balance while performing functional tasks. Each item is scored between 0 and 4. Balance is considered good if the total score is 45 and above.
Dynamic Gait Index | First day
  It consists of 8 walking activities: normal walking, fast-slow walking, walking with horizontal and vertical head movements, walking by jumping from the disabled floor and walking around the obstacle, and turning 360 degrees abruptly on command, going up and down the stairs. During these 8 activities, the patient's performance is scored between 0-3 (0=severe, 3=normal) and the total score is recorded.
Activity-Specific Balance Confidence Scale | First day
  It is a scale that evaluates how confidently people can do 16 activities outside and inside the home. Activities are scored between 0 (unsafe) and 100 (completely confident). A score is obtained by dividing the total score by 16. A higher score indicates greater confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Kahramanmaras Sutcu Imam University